CLINICAL TRIAL: NCT01056042
Title: Postoperative Intramuscular Depot Medroxyprogesterone Acetate Versus Continuous Oral Contraceptive for Pelvic Pain Associated With Endometriosis : Randomized Comparative Trial.
Brief Title: Efficacy of Injectable Contraceptive and Oral Contraceptive Administered After Surgical Treatment of Endometriosis With Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sopon Cheewadhanaraks, Associate Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 50/370-029
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Endometriosis
Keywords: pelvic pain; postoperative; medical therapy
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Intramuscular depot medroxyprogesterone acetate
  Interventions: Drug: intramuscular depot medroxyprogesterone acetate
- B (Active Comparator): ethinyl estradiol 30 micrograms combined with gestodene 75 micrograms
  Interventions: Drug: ethinyl estradiol 30 micrograms, gestodene 75 micrograms

INTERVENTIONS:
Drug: intramuscular depot medroxyprogesterone acetate — 150 mg, Intramuscular, every 3 months
  Other Names: Depo Provera
  Arms: A
Drug: ethinyl estradiol 30 micrograms, gestodene 75 micrograms — one tablet orally, everyday
  Other Names: Gynera
  Arms: B

SUMMARY:
Patients with endometriosis-associated pain have conservative surgery performed to remove all visible lesions. Then, patients are randomized into two groups. In the first group patients have depot medroxyprogesterone acetate injections every 3 months for a total of 6 months.In the second group patients have oral contraceptive combined pills everyday for 6 months. Patients are followed up on recurrence of pain for 1 year after medication.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women from 18 to 45 years of age with endometriosis-associated pain for at least 6 months who had conservative surgery performed.

Exclusion Criteria:

* Medical therapies for endometriosis other than NSAID within previous 6 months
* Contraindication to the drugs
* Wish to conceive
* Request for extirpative surgery
* Other pelvic pathology ( adenomyosis, chronic PID, submucous myoma uteri )

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Patients' satisfaction with the treatment | 1 year and 6 months

SECONDARY OUTCOMES:
pain reduction and adverse side effects | 1 year and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sopon Cheewadhanaraks, M.D., Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Background] Vercellini P, Frontino G, De Giorgi O, Pietropaolo G, Pasin R, Crosignani PG. Continuous use of an oral contraceptive for endometriosis-associated recurrent dysmenorrhea that does not respond to a cyclic pill regimen. Fertil Steril. 2003 Sep;80(3):560-3. doi: 10.1016/s0015-0282(03)00794-5. PMID 12969698
- See also: Faculty of Medicine, Prince of Songkla University — http://medinfo.psu.ac.th